CLINICAL TRIAL: NCT04497207
Title: Classification of Color-Coded Scheimpflug Camera Corneal Tomography Images Using Deep Learning
Brief Title: Deep Learning for Classification of Scheimpflug Corneal Tomography Images
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate professor of Ophthalmology, Assiut University
Other Study IDs: 17300437
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Eye Diseases
Keywords: Keratoconus; Deep learning; Scheimpflug camera; Corneal tomography
MeSH Terms: conditions — Eye Diseases; Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Keratoconus: Those with a clinical diagnosis of keratoconus such as:
  a) the presence of a central protrusion of the cornea with Fleischer ring, Vogt striae, or both by slitlamp examination.(b) an irregular cornea determined by distorted keratometry mires and distortion of retinoscopic red reflex or both in addition to the following topographic findings as summarized by Pińero and colleagues: focal steepening located in a zone of protrusion surrounded by concentrically decreasing power zones, focal areas with dioptric (D) values >47.0D, inferior- superior(I-S) asymmetry measured to be > 1.4 D or angling of the hemimeridians in an asymmetric or broken bowtie pattern with skewing of the steepest radial axis (SRAX) 2.
  Interventions: Other: Scheimpflug Camera Corneal Tomography
- Subclinical keratoconus: Defined as subtle corneal tomographic changes as the aforementioned keratoconus abnormalities in the absence of slit- lamp or visual acuity changes typical of keratoconus (subclinical keratoconus).
  Interventions: Other: Scheimpflug Camera Corneal Tomography
- Normal: This group comprised refractive surgery candidates and subjects applying for a contact lens fitting with a refractive error of less than 8.0 D sphere with less than 3.0 D of astigmatism and without clinical, topographic or tomographic signs of keratoconus nor suspected keratoconus.
  Interventions: Other: Scheimpflug Camera Corneal Tomography

INTERVENTIONS:
Other: Scheimpflug Camera Corneal Tomography — Pentacam Sheimpflug system(Pentacam HR, Oculus Optikgeräte GmbH, software V.1.15r4 n7) is used for imaging of the anterir and posterior surfaces of the cornea to obtain corneal tomographic maps.

SUMMARY:
Keratoconus is a common disorder. An early diagnosis influences the disease prognosis in the affected patients and prevents postoperative complications in patients with keratoconus considering refractive surgery. Machine learning approaches have been widely used for image classification. Here, we will assess the ability of deep learning to enable high-performance image classification of the color-coded corneal maps obtained by Scheimpflug camera in patients with keratoconus, subclinical keratoconus, and normal individuals.

ELIGIBILITY:
Inclusion Criteria:

Keratoconus group:

* Presence of a central protrusion of the cornea with Fleischer ring, Vogt striae, or both by slitlamp examination.
* irregular cornea determined by distorted keratometry mires and distortion of retinoscopic red reflex or both in addition to the following topographic findings as summarized by Pińero and colleagues :
* focal steepening located in a zone of protrusion surrounded by concentrically decreasing power zones
* focal areas with diopteric (D) values >47.0D
* inferior- superior(I-S) asymmetry measured to be > 1.4 D
* Angling of the hemimeridians in an asymmetric or broken bowtie pattern with skewing of the steepest radial axis(SRAX) .

Suspicious group:

• Defined as subtle corneal tomographic changes as the aforementioned keratoconus abnormalities in the absence of slit- lamp or visual acuity changes typical of keratoconus (forme fruste keratoconus).

Normal group:

* Refractive surgery candidates
* Refractive error of less than 8.0 D sphere
* Less than 3.0 D of astigmatism
* without clinical, topographic or tomographic signs of keratoconus or suspect keratoconus.

Exclusion Criteria:

* Systemic disease
* Other corneal disease such as pellucid marginal degeneration
* History of trauma
* Corneal surgery such as corneal cross- linking for progressive keratoconus.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with keratoconus, subclinical keratoconus & normal individuals from refractive surgery candidates.
Sampling Method: Probability Sample
Enrollment: 1669 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Croppedm denoised, and resized to obtain four separate image stacks of 256×256 pixels | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No